CLINICAL TRIAL: NCT02495805
Title: Ultrasound-guided Continuous Proximal Adductor Canal Versus Continuous Femoral Nerve Block for Postoperative Pain Control and Rehabilitation Following Total Knee Arthroplasty
Brief Title: Ultrasound-guided Continuous Proximal Adductor Canal vs Continuous Femoral Nerve Block for Postoperative Pain Control and Rehabilitation Following Total Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never officially began- currently closed with IRB.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1508016335
Record Dates: First submitted 2015-06-30; First posted 2015-07-13 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Total Knee Arthroplasty
Keywords: a continuous proximal adductor canal block (ACB); continuous femoral nerve block (FNB)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adductor canal block (ACB) (Active Comparator): Subjects randomized to this groups receive a continuous proximal adductor canal block (ACB) during surgery.
  Interventions: Procedure: Continuous proximal adductor canal block
- femoral nerve block (FNB) (Active Comparator): Subjects randomized to this groups receive a continuous femoral nerve block (FNB) during surgery.
  Interventions: Procedure: Continuous femoral nerve block

INTERVENTIONS:
Procedure: Continuous proximal adductor canal block — Subjects will be randomized into 2 groups: those who will receive a continuous proximal adductor canal block (ACB) and those who will receive a continuous femoral nerve block (FNB).
  Other Names: ACB
  Arms: adductor canal block (ACB)
Procedure: Continuous femoral nerve block — Subjects will be randomized into 2 groups: those who will receive a continuous proximal adductor canal block (ACB) and those who will receive a continuous femoral nerve block (FNB).
  Other Names: FNB
  Arms: femoral nerve block (FNB)

SUMMARY:
The purpose of the study is to compare continuous femoral nerve block with continuous proximal adductor canal block for postoperative pain control and rehabilitation.

DETAILED DESCRIPTION:
Patients meeting the criteria: American Society of Anesthesiologists (ASA) class I and II, that are scheduled for elective total knee arthroplasty, will be recruited into the study. Subjects will be randomized into 2 groups: those who will receive a continuous proximal adductor canal block (ACB) and those who will receive a continuous femoral nerve block (FNB).

ELIGIBILITY:
Inclusion Criteria:

* Patients with an American Society of Anesthesiologists Physical Status Classification System (ASA) score of 1 or 2 that are healthy without systemic disease or have mild systemic disease, respectively.
* The patient will need to be able to have decision-making capacity and ability to consent for the study.

Exclusion Criteria:

* Patients with an American Society of Anesthesiologists Physical Status Classification System (ASA) score greater than 2.
* Patients unable to have decision-making capacity and ability to consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Motor effects | 24 hours (postoperatively)
  Subjects' change in motor effects will be assessed as maximum voluntary isometric contraction (MVIC) in the quadriceps muscle.

SECONDARY OUTCOMES:
Pain score | On average between 6 and 8 hours postoperatively
  Subjects' pain will be assessed using a numerical pain score, where 10 is the greatest amount of pain.
Pain score | 24 hours (postoperatively)
  Subjects' pain will be assessed using a numerical pain score, where 10 is the greatest amount of pain.
Opioid consumption | On average between 6 and 8 hours postoperatively
  Subjects' pain will be assessed by tracking opioid consumption postoperatively.
Opioid consumption | 24 hours (postoperatively)
  Subjects' pain will be assessed by tracking opioid consumption postoperatively.
Motor effects | On average between 6 and 8 hours postoperatively
  Subjects' change in motor effects will be assessed as maximum voluntary isometric contraction (MVIC) in the quadriceps muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Richa Wardham, MD, Principal Investigator — Yale University